CLINICAL TRIAL: NCT03040739
Title: Treatment of Acetabulum Fracture With O'ARM Surgical Imaging
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: COTYLE_O'ARM
Record Dates: First submitted 2017-01-31; First posted 2017-02-02 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Acetabulum Fracture
Keywords: O'ARM

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case
  Interventions: Other: use of O'ARM imaging system
- control
  Interventions: Other: use of O'ARM imaging system

INTERVENTIONS:
Other: use of O'ARM imaging system — use of O'ARM imaging system

SUMMARY:
Acetabulum fracture are high energy trauma in young people as it can be the result of a simple fall in elder people. This fracture generates an incongruity between acetabulum and femoral head. So surgery is recognized as the best treatment even if technically difficult because of the the complexity of anatomy.Navigation is widely used in orthopaedic surgery .

The aim of the study is to evaluate the effect of peroperative navigation system on reduction of the acetabulum articular surface

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* acetabulum fracture dating less than a month

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patients admitted in the service of orthopaedic surgery for fracture of the cotyle
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Height of incongruity | Day 1
  Reduction of the articular surface of the acetabulum

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided